CLINICAL TRIAL: NCT03057860
Title: TREATgermany: German National Clinical Registry: Treatment and Medical Care of Patients With Moderate-to-severe Atopic Dermatitis
Brief Title: TREATgermany: German National Clinical Registry for Patients With Moderate-to-severe Atopic Dermatitis
Acronym: TREATgermany
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: EK-118032016
Record Dates: First submitted 2017-02-07; First posted 2017-02-20 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Moderate-to-severe Atopic Dermatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No study intervention

SUMMARY:
About 60% of all patients with AD are adults. However, the prevalence and incidence is significantly higher in childhood and adolescence.

Some children, adolescents and adults with moderate-to-severe AD cannot be sufficiently controlled with topical treatments alone and require intermittent or continuous treatment with systemic immunomodulating agents or UV-therapy.

Systematic reviews indicate that although several different interventions for moderate-to-severe AD have been studied in clinical trials, strong recommendations are only possible for Dupilumab in adults and the short-term use of cyclosporin A (CSA).

Pharmaceutical treatment of patients suffering from AE is diverse and frequently not in line with the current guidelines (for example S2-guideline in Germany).

Large head-to-head trials are missing so that long-term effectiveness of systemic interventions for moderate-to-severe AD is speculative.

In this situation, clinical registries can provide valuable information for evidence-based clinical decision making.

Extension of TREATgermany to children and adolescents is necessary as

* moderate-to-severe AD is frequent in this age group, but the effectiveness of existing topical and systemic agents in the routine care setting on clinical severity, patient-reported outcomes, and the course of AD and associated atopic and non-atopic comorbidities over time is still poorly understood
* it is unclear how many children and adolescents cannot be effectively controlled with the avoidance of trigger factors, patient education, and topical anti-inflammatory treatment alone
* innovative agents will become available for these age groups within the next years and reference data will be necessary to evaluate their effectiveness and indication criteria
* adequate evidence regarding patient needs in children and adolescents with moderate-to-severe AD is urgently needed to provide value-based healthcare for this vulnerable patient group
* Best-practice models of transition from adolescent to adult care of patients with moderate-to-severe AD do not exist yet, but constitute a prerequisite for the establishment of efficient patient care

DETAILED DESCRIPTION:
Study procedures:

No study related intervention will be performed. Included patients will be prospectively followed for at least 24 months. A maximum duration of follow-up is not intended.

During the observation period standardized study visits are performed to prospectively document patient characteristics, clinical data, patient-reported outcomes, physician's reasons for treatment decisions, and satisfaction with treatment.

The first study visit is scheduled at patient inclusion (baseline-visit; V1). The second and third study visits are scheduled 3 and 6 months after baseline, respectively. (V2 after 3 months, V3 after 6 months). Thereafter, study visits are scheduled after 3 months (if a new systemic treatment was initiated) or after 6 months (in case no new systemic treatment was prescribed).

In a subset of patients biosamples for molecular analyses including blood, swabs and stool will be taken at baseline and at V6, as well as skin biopsies prior to and 3 months after systemic therapy initiation. This optional module requires separate patient information and informed consent.

Data assessment:

Prospective electronic documentation of disease course and severity, medical care and pharmaceutical treatment of AD.

Pseudomized data will be stored at the registry center (Center for Evidence-based Healthcare, Dresden).

Study assessments include:

1. A short physician report form to document patient history and clinical parameters such as the objective severity of clinical signs, affected body regions, physician's global assessment of disease severity, course of disease and medical treatment of AD including adverse events.
2. A patient report form to assess important subjective parameters, patient reported outcomes such as symptoms, quality of life, treatment satisfaction, patient's assessment of global disease severity, totally/partial well-controlled weeks.

ELIGIBILITY:
Inclusion Criteria:

* AD according to the United Kingdom (UK) working party diagnostic criteria
* Moderate to severe AD
* Objective SCORAD > 20 or Currently anti-inflammatory systemic treatment for AD or Previous anti-inflammatory systemic treatment for AD within past 24 months

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with moderate-to-severe atopic dermatitis
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Score of Atopic Dermatitis (oSCORAD) | Change from Baseline oSCORAD at 2 years
  Severity scoring of atopic dermatitis: the SCORAD index. Consensus Report of the European Task Force on Atopic Dermatitis: Dermatology 1993;186:23-31

SECONDARY OUTCOMES:
Patient Oriented Eczema Measure (POEM) | Baseline (month 0) - 3 months - 6 months - 12 months - 18 months - 2 years
  Charman CR, Venn AJ, Williams HC: The patient-oriented eczema measure: development and initial validation of a new tool for measuring atopic eczema severity from the patients' perspective. Arch Dermatol 2004;140:1513-1519.
Severity of Pruritus and Sleeping Problems (VAS) | Baseline (month 0) - 3 months - 6 months - 12 months - 18 months - 2 years
  Charman CR, Venn AJ, Williams HC: The patient-oriented eczema measure: development and initial validation of a new tool for measuring atopic eczema severity from the patients' perspective. Arch Dermatol 2004;140:1513-1519.
Flares (totally/well controlled weeks) | Baseline (month 0) - 3 months - 6 months - 12 months - 18 months - 2 years
  Schmitt J, Langan S, Deckert S, Svensson A, von KL, Thomas K, Spuls P: Assessment of clinical signs of atopic dermatitis: A systematic review and recommendation. J Allergy Clin Immunol 2013;10.
Health-related Quality of Life (DLQI) | Baseline (month 0) - 3 months - 6 months - 12 months - 18 months - 2 years
  Finlay AY, Khan GK: Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol 1994;19:210-216.
Eczema Area and Severity Index (EASI) | Baseline (month 0) - 3 months - 6 months - 12 months - 18 months - 2 years
  Hanifin JM, Thurston M, Omoto M, Cherill R, Tofte SJ, Graeber M: The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. EASI Evaluator Group. Exp Dermatol 2001;10:11-18.

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Schmitt, Prof.Dr., Principal Investigator — Center for Evidence-based Healthcare, Technical University Dresden
Locations (3):
- Germany (3):
  - Clinics for Dermatology, Allergy and Venerology, Hannover Medical School, Hanover, Lower Saxony
  - Department of Dermatology, UniversityAllergyCenter, Medical Faculty Carl Gustav Carus, TU Dresden, Dresden, Saxony
  - Head Centre for Inflammatory Skin Diseases, Department of Dermatology and Allergy, University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: All Information about the Register-Project — http://www.treatgermany.org

DOCUMENTS (1):
  • Study Protocol (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT03057860/Prot_000.pdf